CLINICAL TRIAL: NCT03739359
Title: Investigating the Role of Gas Flow in Transnasal Pulmonary Aerosol Delivery Via Nasal Cannula: A Double-blinded, Randomized Controlled Trial
Brief Title: The Role of Gas Flow in Transnasal Pulmonary Aerosol Delivery: A Double-blinded, Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: People's Liberation Army General Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HFNC-PFT-002
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: COPD Asthma
Keywords: Nasal cannula; Aerosol therapy; Gas flow

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Nebulization will be offered in a one room and pulmonary function test will be performed in the other room. Both patients and the pulmonary function test technician will be masked to the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Gas flow 50 L/min (Active Comparator): In this group, nasal cannula gas flow will be set at 50 L/min.
  Interventions: Other: nasal cannula gas flow
- GF:IF=1 (Experimental): In this group, nasal cannula gas flow will be set at each individual patient's own inspiratory flow (GF:IF=1)
  Interventions: Other: nasal cannula gas flow
- GF:IF=0.5 (Experimental): In this group, nasal cannula gas flow will be set at 50% of each individual patient's own inspiratory flow (GF:IF=0.5)
  Interventions: Other: nasal cannula gas flow

INTERVENTIONS:
Other: nasal cannula gas flow — High flow nasal cannula (HFNC) is a relatively new oxygen device, which provides warmed and humidified oxygen for patients. When patients need to inhale aerosolized medication during HFNC, the nebulizer will be placed in-line in order to provide both treatments. This study will investigate the influence of three flow settings (50 L/min, GF:IF=1, GF:IF=0.5) on the clinical effects of nebulization.

SUMMARY:
Aerosol delivery via nasal cannula has gained increasing popularity, due to its combined benefits from aerosolized medication and heated warm oxygen therapy. In our previous in vitro study, we investigated the effects of the ratio of nasal cannula gas flow to subject's peak inspiratory flow (GF: IF) on the aerosol lung deposition, and we found that aerosol deposition in lung increased as the GF: IF decreased with an optimal GF: IF between 0.1 to 0.5 producing a stable "lung" deposition in both quiet and distress breathing. Thus we aimed to further validate such an optimal GF: IF in patients with reversible airflow limitations by the delivery of bronchodilators. Adult COPD or asthma patients who met ATS/ERS criteria for bronchodilator response in pulmonary function lab will be recruited and consented. After a washout period (1-3 days), patients will receive an escalating doubling dosage (0.5, 1, 2, and 4mg) of albuterol in total volume of 2mL, delivered by mesh nebulizer via nasal cannula. Patients will be randomly assigned to inhale bronchodilator into 3 group using different flows: 50 L/min,GF: IF = 1.0, and GF: IF = 0.5.

DETAILED DESCRIPTION:
Introduction Both in vitro and in vivo radiolabeled studies on nebulization via high flow nasal cannula (HFNC) showed that aerosol lung deposition decreased with the increasing nasal cannula gas flow, which, however, was not observed in patients with distressed breathing. In our previous in vitro study, we investigated the effects of the ratio of nasal cannula gas flow to subject's peak inspiratory flow (GF: IF) on the aerosol lung deposition, and we found that aerosol deposition in lung increased as the GF: IF decreased with an optimal GF: IF between 0.1 to 0.5 producing a stable "lung" deposition in both quiet and distress breathing. Thus we aimed to further validate such an optimal GF: IF in patients with reversible airflow limitations by the delivery of bronchodilators.

Methods and analysis COPD and asthma patients with positive response to four actuations of albuterol via metered dose inhaler (MDI) and valved holding chamber (VHC) will be enrolled and consented in the study. After a washout period (1-3 days), patients will be randomly assigned to three groups with different nasal cannula gas flow: 50L/min, GF: IF = 1.0, and GF: IF = 0.5. In each treatment arm, patients will firstly receive saline, then followed by an escalating doubling dosages (0.5, 1, 2, and 4mg) of albuterol in a total volume of 2mL, delivered by mesh nebulizer (VMN, Aerogen, Ireland) via heated nasal cannula at 37℃. An interval of 30 min will be maintained between two doses of albuterol, and pulmonary spirometry will be measured at baseline and after each dose. Titration will be terminated when an additional FEV1 improvement was < 5%.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with positive bronchodilator responses to four actuations of albuterol (Ventolin, GSK, UK) via MDI with VHC (OptiChamber Diamond, Philips, USA) will be eligible for enrollment. A positive bronchodilator response is defined in accordance with ATS/ERS guidelines as follows: an increase in FEV1 of ≥ 12% and absolute change ≥ 200 mL from baseline.

Exclusion Criteria:

* age ≥ 90 years old;
* pregnancy;
* pulmonary exacerbation within two weeks before enrollment;
* reluctant to participate;
* inability to complete the follow-up spirometry after each bronchodilator inhalation;
* resting heart rate > 100bpm;
* resting systolic blood pressure > 160mmHg or diastolic blood pressure > 110mmHg.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
The number of patients who meet the positive criteria of responding to albuterol at the dose of 0.5mg | 30 minutes
  The number of patients in HFNC nebulization who respond to albuterol at the dose of 0.5mg
The number of patients who meet the positive criteria of responding to albuterol at the dose of 1.5 mg | 60 minutes
  The number of patients in HFNC nebulization who respond to albuterol at the dose of 1.5mg
The number of patients who meet the positive criteria of responding to albuterol at the dose of 3.5 mg | 90 minutes
  The number of patients in HFNC nebulization who respond to albuterol at the dose of 3.5mg
The number of patients who meet the positive criteria of responding to albuterol at the dose of 7.5mg | 120 minutes
  The number of patients in HFNC nebulization who respond to albuterol at the dose of 7.5mg

SECONDARY OUTCOMES:
the accumulative dose of albuterol required across groups to produce positive bronchodilation effects | 120 minutes
  the accumulative dose of albuterol required to produce positive bronchodilation effects in each group
the incidence of side effect (tachycardia) in each group | 120 minutes
  the incidence of side effect (tachycardia) will be recorded in each group
the incidence of side effect (tremor) in each group | 120 minutes
  the incidence of side effect (tachycardia) will be recorded in each group

CONTACTS AND LOCATIONS:
Overall Officials: Lixing Xie, MD, Study Chair — People's Liberation Army General Hospital
Locations (1):
- People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after deidentification that underlie the reports reported in this article can be obtained by contacting the corresponding author. Data will be available immediately following publication and ending in 5 years.
Supporting Information: Study Protocol
Time Frame: 5 years following publication
Access Criteria: contacting the corresponding author

REFERENCES:
- [Result] Zhu Y, Yin H, Zhang R, Wei J. High-flow nasal cannula oxygen therapy versus conventional oxygen therapy in patients with acute respiratory failure: a systematic review and meta-analysis of randomized controlled trials. BMC Pulm Med. 2017 Dec 13;17(1):201. doi: 10.1186/s12890-017-0525-0. PMID 29237436
- [Result] Braunlich J, Wirtz H. Oral Versus Nasal High-Flow Bronchodilator Inhalation in Chronic Obstructive Pulmonary Disease. J Aerosol Med Pulm Drug Deliv. 2018 Aug;31(4):248-254. doi: 10.1089/jamp.2017.1432. Epub 2017 Dec 20. PMID 29261402
- [Result] Gacouin A, Maamar A, Fillatre P, Sylvestre E, Dolan M, Le Tulzo Y, Tadie JM. Patients with preexisting psychiatric disorders admitted to ICU: a descriptive and retrospective cohort study. Ann Intensive Care. 2017 Dec;7(1):1. doi: 10.1186/s13613-016-0221-x. Epub 2017 Jan 3. PMID 28050894
- [Result] Ammar MA, Sasidhar M, Lam SW. Inhaled Epoprostenol Through Noninvasive Routes of Ventilator Support Systems. Ann Pharmacother. 2018 Dec;52(12):1173-1181. doi: 10.1177/1060028018782209. Epub 2018 Jun 12. PMID 29890848
- [Result] Dugernier J, Hesse M, Jumetz T, Bialais E, Roeseler J, Depoortere V, Michotte JB, Wittebole X, Ehrmann S, Laterre PF, Jamar F, Reychler G. Aerosol Delivery with Two Nebulizers Through High-Flow Nasal Cannula: A Randomized Cross-Over Single-Photon Emission Computed Tomography-Computed Tomography Study. J Aerosol Med Pulm Drug Deliv. 2017 Oct;30(5):349-358. doi: 10.1089/jamp.2017.1366. Epub 2017 May 2. PMID 28463044
- [Derived] Li J, Luo J, Chen Y, Xie L, Fink JB. Effects of flow rate on transnasal pulmonary aerosol delivery of bronchodilators via high-flow nasal cannula for patients with COPD and asthma: protocol for a randomised controlled trial. BMJ Open. 2019 Jun 24;9(6):e028584. doi: 10.1136/bmjopen-2018-028584. PMID 31239304